CLINICAL TRIAL: NCT02058030
Title: The 3 cm of Head Elevation Provides Higher Insertion Success Than do the 6 cm of it for ProSeal Laryngeal Mask Airway Insertion in Adult Patients
Brief Title: The Influence of Degree of Head Elevation on Insertion Success for ProSeal Laryngeal Mask Airway Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Center, Seoul (Other)
Responsible Party: Principal Investigator, Sung Hoon Kim, MD, National Medical Center, Seoul
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: phdkim1
Record Dates: First submitted 2013-10-08; First posted 2014-02-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia
Keywords: ProSeal laryngeal mask airway; Insertion success; complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3cm head elevation (Other): Insertion of ProSeal laryngeal mask airway
  Interventions: Device: Insertion of ProSeal laryngeal mask airway
- 6cm head elevation (Active Comparator): Insertion of ProSeal laryngeal mask airway
  Interventions: Device: Insertion of ProSeal laryngeal mask airway

INTERVENTIONS:
Device: Insertion of ProSeal laryngeal mask airway — The patient's head was placed on the 3 cm or 6 cm height of a pillow in supine and PLMA was inserted using a standard method in the sniffing position.
  The success rate at first and second attempt, insertion time, Seal pressure, hemodynamic variables, complications(blood staining on cuff, sore throat and hoarseness) were assessed

SUMMARY:
Background - The purpose of the present study is to evaluate the success and pharyngeal trauma when 3 or 6 cm height of pillow is used for the ProSealTM laryngeal mask airway insertion

Methods

- This prospective randomized, controlled study included 80 adult patients . In the 3 cm (n=40) or 6 cm group (n=40), the PLMA was inserted while the head is placed on the 3 cm or 6 cm height of pillow. The success rate at first and second attempt, insertion time, blood staining on cuff, sore throat and hoarseness were assessed.

DETAILED DESCRIPTION:
Background: The "sniffing position" (i.e., the neck flexed and head extended by means of a pillow) eases tracheal intubation because the three axes, namely, the axis of the mouth, the pharyngeal axis and the laryngeal axis, are put in almost a straight line. The benefit of the sniffing position that align three axis could possibly be applicable when the ProSeal LMA is inserted. For the endotracheal intubation, it has been recommended to elevate the patient's head 8 to 10 cm with pads under the occiput (shoulder remaining on the table) and extend the head at the atlanto-occipital joint to align the oral, pharyngeal, and laryngeal axes such that the passage and line of vision from the lips to the glottic opening are most nearly a straight line.

There have been several clinical studies about the effect of head and neck position including neutral, flexion or extension on the ease of LMA insertion.

However, it has not been much recommended or investigated about the influence of head elevation on the insertion success of PLMA until now. The purpose of the present study is to evaluate the success and pharyngeal trauma when 3 or 6 cm height of pillow is used for the ProSeal laryngeal mask airway insertion in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-2
* scheduled for minor surgery in the supine position were enrolled

Exclusion Criteria:

* cardiorespiratory disease patients
* patients were at risk of aspiration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
insertion success rate | 2013.11 - 2014.12

SECONDARY OUTCOMES:
complication | 2013.11- 2014.12
  Number of participants with blood on the surface of the cuff, postoperative sore throat and hoarseness as indices of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mija Yun, MD, PhD, Study Chair — National medical center
Locations (1):
- National Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Yun MJ, Hwang JW, Kim SH, Hong HJ, Jeon YT, Park HP. Head elevation by 3 vs. 6 cm in ProSeal laryngeal mask airway insertion: a randomized controlled trial. BMC Anesthesiol. 2016 Aug 5;16(1):57. doi: 10.1186/s12871-016-0220-3. PMID 27494933